CLINICAL TRIAL: NCT00233428
Title: Phase 1 Study to Determine Racial and Gender Differences in Platelet Aggregation
Brief Title: Study to Determine Racial and Gender Differences in Platelet Aggregation
Status: Completed | Type: Observational
Sponsor: Texas Tech University Health Sciences Center (Other)
Other Study IDs: L05-108
Record Dates: First submitted 2005-10-03; First posted 2005-10-05 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-05

CONDITIONS: Platelet Aggregation
Keywords: Healthy volunteers
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective

INTERVENTIONS:
Procedure: Blood Draw

SUMMARY:
The purpose of this study is to see if there is a racial and/or gender difference in platelet aggregation.

DETAILED DESCRIPTION:
Genetic variability of various components of the coagulation system has been reported. Data on racial and gender differences in platelet aggregation are lacking.

We hypothesize that there are significant racial and gender differences on aggregatory response of platelets to commonly used agonists to evaluate platelet function such as adenosine diphosphate (ADP), epinephrine, collagen and arachidonic acid.

ELIGIBILITY:
Inclusion Criteria:

* Race of Caucasian, African American, or Hispanic

Exclusion Criteria:

* Chronic medical conditions
* Tobacco use
* Regular non-steroidal anti-inflammatory use, aspirin use, or use of one of the other anti-platelet drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-05; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chanwit Roongsritong, MD, Principal Investigator — TTUHSC
Locations (1):
- TTUHSC, Lubbock, Texas, United States

REFERENCES:
- [Derived] Otahbachi M, Simoni J, Simoni G, Moeller JF, Cevik C, Meyerrose GE, Roongsritong C. Gender differences in platelet aggregation in healthy individuals. J Thromb Thrombolysis. 2010 Aug;30(2):184-91. doi: 10.1007/s11239-009-0436-x. PMID 20039102